CLINICAL TRIAL: NCT06149156
Title: Efficacy of a Mobile Health Mindfulness-based Intervention on Resident Well-being and Performance
Brief Title: Resident Well-being and Performance
Acronym: ResiWell
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1432; A171600 (Other: UW Madison); IRB Approval 2/9/2024 (Other: UW Madison)
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Burnout, Psychological
Keywords: Residency; Well-being; Physician Health; Physician Burnout; Mindfulness; Mobile health
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Minds Program (HMP) intervention (Experimental): Participants will receive access to the 4-week HMP Foundations module. The HMP app is a meditation-based smartphone app designed to promote and protect psychological well-being through sustainable skills training. The program is grounded in constituents of psychological well-being identified in empirical literature. HMP provides core content, with instruction administered through a curriculum of guided practices. HMP is based on research on eudaimonic well-being (e.g., environmental mastery, purpose) and brain-based skills that underlie these qualities (e.g., regulation of attention, mental flexibility). The full HMP has guided audio practices that address 4 constituents of well-being: awareness, connection, insight, and purpose. At post-treatment, participants will be given access to additional HMP content to support their continued practice.
  Interventions: Behavioral: Healthy Minds Program App
- Waitlist Control (Active Comparator): Participants will receive a list of well-being resources. They will be given access to HMP at the end of the study.
  Interventions: Behavioral: Well-being Resources

INTERVENTIONS:
Behavioral: Healthy Minds Program App — The four-week intervention comprises two introductory lessons and guided meditations followed by one week of content for each pillar of well-being. Each week includes two brief lessons (5-7 minutes) with education on the scientific research behind the practices, as well as examples of how to strengthen the skills of each pillar in daily life, along with three guided meditations for which the participant can select the practice length (5-30 minutes).
  Arms: Healthy Minds Program (HMP) intervention
Behavioral: Well-being Resources — List of well-being resources that comprises of online video links and books
  Arms: Waitlist Control

SUMMARY:
This project aims to investigate the effectiveness of a meditation intervention utilizing a smart phone-based meditation app on resident burnout, well-being, and performance self-efficacy in a randomized clinical trial. 500 participants will be enrolled for a 4 week intervention.

DETAILED DESCRIPTION:
Burnout is an increasingly prevalent challenge in the medical field and especially prominent in residency. Burnout negatively affects learning and decision-making, physician performance, and patient outcomes. Studies have shown that mindfulness-based interventions are effective at reducing burnout and strengthening well-being in physicians. Furthermore, mobile health mindfulness-based interventions have similar benefits to in-person interventions while offering the advantages of increased scalability, lack of physical constraint, and lower costs. This project will use a novel mobile health MBI and measure resident burnout, well-being, and self-efficacy in performance.

ELIGIBILITY:
Inclusion Criteria:

* Resident in a high burnout rate specialty: family medicine, internal medicine, obstetrics and gynecology, emergency medicine, general surgery, or surgical sub-specialty (plastic surgery, urology, neurosurgery, orthopedic surgery, vascular surgery, cardiothoracic surgery, otolaryngology, ophthalmology)

Exclusion Criteria:

* Participants who have previously used the HMP (a version of HMP has been freely available to the public since 2020)
* Participants who have been practicing meditation daily or almost daily for the prior six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Stress Measured by the Perceived Stress Scale | baseline, week 1, week 2, week 3, week 4, 3 months
  The Perceived Stress Scale is a 10-item scale where participants report their level of perceived stress (e.g., "In the last week, how often have you felt nervous and 'stressed'?"). It is scored on a 5-point Likert scale where 0 = "never" to 4 = "very often." Total scores range from 0 to 40 where higher scores indicate greater perceived stress.

SECONDARY OUTCOMES:
Change in Burnout Measured by the Abbreviated Maslach Burnout Inventory: Personal Accomplishment Dimension | baseline, 4 weeks, 3 months
  The Abbreviated Maslach Burnout Inventory (MBI) is a 9-item questionnaire to assesses burnout as a continuum on three different dimensions: Emotional Exhaustion, Depersonalization, and reduced Personal Accomplishment. It is scored on a 6-point Likert scale. Total possible range of scores for each sub-scale is 0-18, lower scores on the Personal Accomplishment dimension indicate higher burnout..
Change in Burnout Measured by the Abbreviated Maslach Burnout Inventory: Depersonalization and Emotional Exhaustion Dimensions | baseline, 4 weeks, 3 months
  The Abbreviated Maslach Burnout Inventory (MBI) is a 9-item questionnaire to assesses burnout as a continuum on three different dimensions: Emotional Exhaustion, Depersonalization, and reduced Personal Accomplishment. It is scored on a 6-point Likert scale. Total possible range of scores for each sub-scale is 0-18, higher scores on the Depersonalization and Emotional Exhaustion dimensions indicate higher burnout.
Change in Flourishing Measured by the Flourishing Index Score | baseline, 4 weeks, 3 months
  The Flourishing Index is a 10-item questionnaire where participants report their general level of flourishing (e.g., well-being, health, etc.). It is scored on a 0 to 10-point scale, with anchors varying across items. The total score ranges from 0 to 100 with higher scores indicating higher flourishing.
Change in Resilience Measured by the Brief Resilience SCale | baseline, 4 weeks, 3 months
  The Brief Resilience Scale is a 6-item questionnaire where participants report their resilience in responding to difficult events or setbacks. It is scored on a 0-6 scale, with the total score being the average of scores across all items with higher scores indicating higher resilience.
Change in Sleep Disturbance Measured by Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Score | baseline, 4 weeks, 3 months
  The PROMIS Sleep Disturbance scale is a computer-adaptive measure where participants report how often in the past 7 days they had various sleep-related experiences (e.g., "my sleep was restful"). It is scored on a 5-point Likert scale where 1 = not at all to 5 = very much. It provides total scores as T-scores (mean = 50, standard deviation (SD) = 10) where higher scores indicate more sleep disturbance.
Change in Awareness Measured by Five Facet Mindfulness Questionnaire Acting with Awareness Subscale Score | baseline, 4 weeks, 3 months
  he Five Facet Mindfulness Questionnaire Acting with Awareness Subscale is a 8-item subscale where participants report on their general ability to focus. It is scored on a 5-point Likert scale where 1 = never or very rarely true to 5 = very often or always true. The total possible range of scores is 8-40 where higher scores indicate a greater ability to focus.
Change in Healthy Minds Index (HM Index) | baseline, week 1, week 2, week 3, week 4, 3 months
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0 to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Scores between 0 and 4 will be reported where higher scores indicate more of each quality.
Change in General Self-Efficacy Measured by the General Self-Efficacy Scale | baseline, 4 weeks, 3 months
  The General Self-Efficacy Scale is a 10-item questionnaire where participants report their general sense of perceived self-efficacy in coping with daily hassles and experiencing stressful life events. It is scored on a 4-point Likert sale and is summed into a total score ranging from 10-40. Higher scores indicate higher general self-efficacy
Change in Self-efficacy of Performance Measured by self-report on Accreditation Council for Graduate Medical Education (ACGME) Residency Milestones | baseline, 4 weeks, 3 months
  The Accreditation Council for Graduate Medical Education Milestones are an assessment of core competencies for residents to track progression. We will assess Milestones in the core competencies of Patient Care, Practice-Based Learning and Improvement, Professionalism, and Interpersonal and Communication Skills. Participants will report their self-assessment of milestones on a 1-5 Likert scale.
Change in Connection Measured by NIH Toolbox Loneliness Score | baseline, 4 weeks, 3 months
  The NIH Toolbox Loneliness is a 5-item questionnaire where participants report how often in the past week they have felt loneliness. It is scored on a 5-point Likert scale where 1 = never to 5 = always. The total possible range of scores is 5-25 where higher scores indicate a greater sense of loneliness.
Change in Meaning in Life Measured by NIH Toolbox Meaning and Purpose Score | baseline, 4 weeks, 3 months
  The PROMIS / NIH Toolbox Meaning and Purpose is a computer-adaptive measure where participants report how much meaning and purpose they experience in life (e.g., "I understand my life's meaning"). It is scored on a 5-point Likert scale where 1 = strongly disagree to 5 = strongly agree. It provides total scores as T-scores (mean = 50, SD = 10) where higher scores indicate more meaning and purpose in life.

OTHER OUTCOMES:
Change in Digital Working Alliance Inventory | 4 weeks
  The Digital Working Alliance Inventory is a 6-item scale where participants report their working alliance with the HMP app (e.g., "The HMP app supports me to overcome challenges"). It is scored on a 7-point Likert scale where 1 = "strongly disagree" to 7 = "strongly agree." Total scores range from 6 to 42 where higher scores indicate greater working alliance.
Acceptability, Appropriateness, and Feasibility of Intervention | 4 weeks
  The Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Outcome Measure (FIM) is a 12-iten scale where participants report their perceived acceptability, appropriateness, and feasibility of the intervention in residency. It is scored on a 5-point Likert scale with total scores as the average for each domain. Higher scores indicated higher acceptability, appropriateness, and feasibility of the measure.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No